CLINICAL TRIAL: NCT03709264
Title: Intravenous Amino Acid Therapy for Kidney Protection in Cardiac Surgery: a Multi-centre Randomized Blinded Placebo Controlled Clinical Trial.
Brief Title: Intravenous Amino Acid Therapy for Kidney Protection in Cardiac Surgery.
Acronym: PROTection
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Università Vita-Salute San Raffaele (Other)
Responsible Party: Principal Investigator, Giovanni Landoni, MD, Associate Professor, Università Vita-Salute San Raffaele
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PROTection/47/OSR
Record Dates: First submitted 2018-10-09; First posted 2018-10-17 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Cardiac Surgery
Keywords: kidney protection; acute kidney injury; cardiac surgery; amino acids; mortality; ICU
MeSH Terms: conditions — Acute Kidney Injury | interventions — Amino Acids

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Amino Acids infusion (Experimental)
  Interventions: Drug: Amino Acids
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Amino Acids — Patients randomized to experimental arm receive a continuous infusion of a balanced mixture of amino acids in a dose of 2 g/kg ideal body weight/day (to a maximum 100 g/day) from the operating room admission up to either death, start of RRT, ICU discharge or 72 hours after treatment initiation, trough a central venous line
  Arms: Amino Acids infusion
Drug: Placebos — Placebo: standard treatment
  Arms: Placebo

SUMMARY:
To date, no pharmacological agents are proven efficacious in treating perioperative AKI. There is a strong biological rationale for the administration of amino acid in the management of patients at risk of AKI with increases in renal blood flow and GFR of 25 to 60% for several hours after the administration of amino acids (Woods LL 1993) mediated by a afferent arteriolar dilation.(Meyer TW 1983) Moreover, animal models have demonstrated that an increase in renal blood flow in response to a short-term amino acid infusion can protect the kidney from acute ischemic insults. Finally, these nephro-protective effects are preserved in critical illness. Cardiac surgery appears to be the best setting to test the likely beneficial renal effects of amino acid because of pathophysiological principles and the ability to intervene before the injury has begun. Although the etiology of AKI in cardiac surgery is multifactorial, renal hypoperfusion is believed to play a major role in this development by decreasing renal perfusion through a reduction in renal blood flow and through the activation of the sympathetic nervous system and the renin-angiotensin system with afferent arteriolar vasoconstriction. In this setting, a global increase in renal blood flow by means of Amino Acid therapy appears a logical and promising intervention.

The primary aim of the study is to determine whether providing continuous infusion of a balanced mixture of amino acids, compared to placebo (balanced crystalloid solution), reduces the incidence of acute kidney injury (AKI) in patients scheduled for cardiac surgery defined as KDIGO stage 1 or greater during hospital stay.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years
* scheduled cardiac surgery
* expected to stay in ICU at least 1 night after surgery
* signed informed consent

Exclusion Criteria:

* Patient currently enrolled into another randomized clinical trial
* Patient currently receiving or scheduled for intermittent or continuous renal replacement therapy
* Patients with CKD of equal or more than CKD stage IV (GFR<30 ml/min/1.73 m2)
* Patient with a kidney transplant
* Patient is not expected to survive ICU or hospital discharge
* Patient previously been enrolled and randomized into this study
* Patient has severe liver disease (Child-Pugh score >7 points)
* Patient has a hypersensitivity (known allergy) to one or more of the included amino acids
* Patient has a congenital alteration of amino acid metabolism
* Pregnant or currently breastfeeding patients
* Patients with any of the contraindications reported in the summary product characteristics.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3511 (Actual)
Dates: Start 2019-10-07 (Actual); Primary Completion 2024-01-17 (Actual); Study Completion 2025-01-17 (Actual)

PRIMARY OUTCOMES:
AKI incidence | Until hospital discharge, an average of 10 days
  Incidence of Acute Kidney Injury during hospital stay

SECONDARY OUTCOMES:
Mortality | 180 days
  All-cause mortality at ICU discharge, hospital discharge, 30 and 90 and 180 days after randomization
RRT | 180 days
  Need and duration of renal replacement therapy
ICU stay | Until ICU discharge, an average of 2 days
  Duration of Intensive Care Unit stay
Hospital stay | Until hospital discharge, an average of 10 days
  Duration of hospital stay
Mechanical Ventilation | Until ICU discharge, an average of 2 days
  Need and duration of mechanical ventilation
EQ-5D | 180 days
  Quality of life at 180 days after randomization as measured by the EQ-5D

CONTACTS AND LOCATIONS:
Locations (22):
- Croatia (2):
  - University Hospital Dubrava, Dubrava
  - Magdalena Clinic for Cardiovascular Diseases, Zagreb
- Italy (19):
  - Ospedale San Carlo, Potenza, Basilicate
  - Ospedale Mater Domini, Catanzaro, Calabria
  - Ospedale Monaldi, Napoli, Campania
  - Pineta Grande Hospital, Castel Volturno, Caserta
  - Azienda Ospedaliera Sant'Andrea, Rome, Lazio
  - Ospedale San Camillo, Rome, Lazio
  - IRCCS San Martino Istitute, Genoa, Liguria
  - IRCCS Cardiologico Monzino, Milan, Lombardy
  - Istituto Clinico Humanitas, Rozzano, Lombardy
  - IRCCS Ospedale San Donato, Miano, Milano
  - Città della Salute, Turin, Piedmont
  - Ospedale Ordine Mauriziano, Turin, Piedmont
  - Maria Cecilia Hospital, Cotignola, Ravenna
  - Ospedale del cuore - Fondazione Toscana Gabriele Monasterio, Massa, Tuscany
  - Ospedale San Raffaele, Milan
  - AOU Policlinico Paolo Giaccone, Palermo
  - Azienda Ospedaliera Universitaria Pisana, Pisa
  - Grande Ospedale Metropolitano, Reggio Calabria
  - Ospedale Santa Maria della Misericordia, Udine
- National University Hospital, Singapore, Singapore

REFERENCES:
- [Background] Losiggio R, Redaelli MB, Landoni G, Bellomo R. Intravenous Amino-acid Infusion to Prevent Acute Kidney Injury after Cardiac Surgery: A Review of the Evidence. Ann Thorac Surg. 2025 Aug;120(2):256-266. doi: 10.1016/j.athoracsur.2024.11.020. Epub 2024 Dec 4. PMID 39643100
- [Background] Baiardo Redaelli M, Landoni G, Monti G, Bellomo R. Amino acids and the kidney; friends or foes? Curr Opin Clin Nutr Metab Care. 2025 Mar 1;28(2):156-159. doi: 10.1097/MCO.0000000000001083. Epub 2024 Oct 21. PMID 39485306
- [Background] Pruna A, Losiggio R, Landoni G, Kotani Y, Redaelli MB, Veneziano M, Lee TC, Zangrillo A, Gaudino MFL, Bellomo R; for Protection Study group. Amino Acid Infusion for Perioperative Functional Renal Protection: A Meta-analysis. J Cardiothorac Vasc Anesth. 2024 Dec;38(12):3076-3085. doi: 10.1053/j.jvca.2024.08.033. Epub 2024 Aug 22. PMID 39384419
- [Background] Landoni G, Brambillasca C, Baiardo Redaelli M, Bradic N, Ti LK, Povsic-Cevra Z, Nepomniashchikh VA, Zoccai GB, D'Ascenzo F, Romagnoli E, Scandroglio AM, Ballotta A, Rondello N, Franco A, Massaro C, Viscido C, Calabro MG, Garofalo E, Canichella F, Monaco F, Severi L, Pisano A, Barucco G, Venditto M, Federici F, Licheri M, Paternoster G, Trompeo A, Belletti A, Mantovani LF, Perone R, Dalessandro G, Kroeller D, Haxhiademi D, Galbiati C, Tripodi VF, Giardina G, Lembo R, Nakhnoukh C, Guarracino F, Longhini F, Bove T, Zangrillo A, Bellomo R, Fominskiy E. Intravenous amino acid therapy for kidney protection in cardiac surgery a protocol for a multi-centre randomized blinded placebo controlled clinical trial. The PROTECTION trial. Contemp Clin Trials. 2022 Oct;121:106898. doi: 10.1016/j.cct.2022.106898. Epub 2022 Aug 28. PMID 36038001
- [Background] Rosario Losiggio, Martina Baiardo Redaelli, Alessandro Pruna, Giovanni Landoni, Rinaldo Bellomo. The renal effects of amino acids infusion. Signa Vitae. 2024. 20(7);1-4.
- [Background] Bellomo R, Monaco F, Paternoster G. Intravenous Amino Acids and Kidney Protection. Reply. N Engl J Med. 2024 Nov 21;391(20):1965-1966. doi: 10.1056/NEJMc2412012. No abstract available. PMID 39566002
- [Background] Kotani Y, Baiardo Redaelli M, Pruna A, Losiggio R, Cocozza S, Ti LK, Bradic N, Comis M, Landoni G, Bellomo R. Intravenous amino acid for kidney protection: current understanding and future perspectives. Clin Kidney J. 2024 Dec 26;18(2):sfae409. doi: 10.1093/ckj/sfae409. eCollection 2025 Feb. PMID 39981140
- [Background] Pruna A, Monaco F, Asiller OO, Delrio S, Yavorovskiy A, Bellomo R, Landoni G. How Would We Prevent Our Own Acute Kidney Injury After Cardiac Surgery? J Cardiothorac Vasc Anesth. 2025 May;39(5):1123-1134. doi: 10.1053/j.jvca.2025.01.019. Epub 2025 Jan 13. PMID 39922732
- [Background] Bottussi A, D'Andria Ursoleo J, Agosta VT, De Luca M, Monaco F. The role of amino acids and protein administration in preventing cardiac surgery-associated acute kidney injury. Future Cardiol. 2025 Mar;21(3):191-202. doi: 10.1080/14796678.2025.2463271. Epub 2025 Feb 8. PMID 39921856
- [Result] Landoni G, Monaco F, Ti LK, Baiardo Redaelli M, Bradic N, Comis M, Kotani Y, Brambillasca C, Garofalo E, Scandroglio AM, Viscido C, Paternoster G, Franco A, Porta S, Ferrod F, Calabro MG, Pisano A, Vendramin I, Barucco G, Federici F, Severi L, Belletti A, Cortegiani A, Bruni A, Galbiati C, Covino A, Baryshnikova E, Giardina G, Venditto M, Kroeller D, Nakhnoukh C, Mantovani L, Silvetti S, Licheri M, Guarracino F, Lobreglio R, Di Prima AL, Fresilli S, Labanca R, Mucchetti M, Lembo R, Losiggio R, Bove T, Ranucci M, Fominskiy E, Longhini F, Zangrillo A, Bellomo R; PROTECTION Study Group. A Randomized Trial of Intravenous Amino Acids for Kidney Protection. N Engl J Med. 2024 Aug 22;391(8):687-698. doi: 10.1056/NEJMoa2403769. Epub 2024 Jun 12. PMID 38865168
- [Result] Baiardo Redaelli M, Monaco F, Bradic N, Scandroglio AM, Ti LK, Belletti A, Viscido C, Licheri M, Guarracino F, Pruna A, Pisano A, Pontillo D, Federici F, Losiggio R, Serena G, Tomasi E, Silvetti S, Ranucci M, Brazzi L, Cortegiani A, Landoni G, Mastroroberto P, Paternoster G, Gaudino MFL, Zangrillo A, Bellomo R; for the PROTECTION Study Group Collaborators. Amino Acid Infusion for Kidney Protection in Cardiac Surgery Patients with Chronic Kidney Disease: A Secondary Analysis of the PROTECTION Trial. Anesthesiology. 2025 May 1;142(5):818-828. doi: 10.1097/ALN.0000000000005336. Epub 2024 Dec 19. PMID 39705670
- [Result] Belletti A, Pisano A, Scandroglio AM, Garofalo E, Calabro MG, Ferrod F, Monaco F, Brambillasca C, Baiardo Redaelli M, Meroi F, Fominskiy E, Vignale R, Ajello S, Venditto M, Scquizzato T, Porta S, Losiggio R, Suriano P, Pontillo D, Orso D, Tomasi E, Paternoster G, Lomivorotov V, Longhini F, Landoni G, Zangrillo A, Maisano F, Bellomo R, Pieri M; PROTECTION Study Group Collaborators. Intravenous amino acids for renal protection in patients receiving temporary mechanical circulatory support: a secondary subgroup analysis of the PROTECTION study. Eur J Cardiothorac Surg. 2025 Feb 4;67(2):ezaf035. doi: 10.1093/ejcts/ezaf035. PMID 39977357
- [Result] Pontillo D, Rong LQ, Pruna A, Pisano A, Monaco F, Bruni A, Baiardo Redaelli M, Ti LK, Belletti A, Bradic N, Massaro C, Barucco G, Viscido C, Losiggio R, Federici F, Marmiere M, Silvetti S, Marchetti C, Carmosino M, Manazza M, Oliva FM, Cortegiani A, Guarracino F, Ranucci M, Paternoster G, Landoni G, Zangrillo A, Gaudino MFL, Bellomo R; PROTECTION Study Group Collaborators. Impact of Cardiopulmonary Bypass Duration on the Renal Effects of Amino Acids Infusion in Cardiac Surgery Patients. J Cardiothorac Vasc Anesth. 2025 Sep;39(9):2296-2306. doi: 10.1053/j.jvca.2025.05.050. Epub 2025 Jun 2. PMID 40571473